CLINICAL TRIAL: NCT04633499
Title: Effects of tDCS on Visual Perspective Taking and Emotion Recognition in Healthy Older Adults
Brief Title: Effects of tDCS on Social Cognition in Aging
Acronym: SoCoStim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: SoCoStim
Record Dates: First submitted 2020-08-27; First posted 2020-11-18 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: Aging; Social Cognition
Keywords: tDCS; Social Cognition
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: It is a randomized, balanced cross-over design with within- as well as between group comparisons. Two groups will be investigate: young participants (n = 30) and older participants (n = 60). The group of young participants will serve as a control group and will only get a neuropsychological assessment of their cognitive abilities at the beginning of the study, an MRI assessment and one session of the investigated paradigms (without tDCS). The group of older participants will conduct a session of MRI assessment and neuropsychological assessment, as well as two tDCS sessions (anodal/sham). The stimulation will either be over the rTPJ or the dmPFC. This set-up is identical to the study of Martin et al., (2020).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will receive either an active or a sham tDCS stimulation. Sham stimulation will use a ramp-up, so that participants are not able to tell whether they are stimulated or not, if they are tDCS naive.
  Sham or active tDCS is applied via codes. Principal Investigators are blinded for these codes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dmPFC tDCS + Social Cognition tasks in older participants (Active Comparator): Participants will receive either active or sham stimulation over the dmPFC while conducting two different social cognition paradigms: one regarding emotion recognition, one on visual perspective taking.
  Interventions: Behavioral: Social Cognition Task; Device: tDCS
- rTPJ tDCS + Social Cognition tasks in older participants (Experimental): Participants will receive either active or sham stimulation over the rTPJ while conducting two different social cognition paradigms: one regarding emotion recognition, one on visual perspective taking.
  Interventions: Behavioral: Social Cognition Task; Device: tDCS
- Social cognition tasks in younger participants (Active Comparator): Participants will conduct two different social cognition paradigms: one regarding emotion recognition, one on visual perspective taking but without tDCS stimulation.
  Interventions: Behavioral: Social Cognition Task

INTERVENTIONS:
Behavioral: Social Cognition Task — Two paradigms will be tested: visual perspective taking and reading the mind in the eyes.
Device: tDCS — tDCS either over the dmPFC or the rTPJ.
  Arms: dmPFC tDCS + Social Cognition tasks in older participants; rTPJ tDCS + Social Cognition tasks in older participants

SUMMARY:
The aim of the study is to explore the effect of transcranial direct current stimulation (tDCS) on either the right tempo-parietal junction (rTPJ) or the dorsomedial prefrontal cortex (dmPFC) in healthy older adults (replication in a different sample of a study by Martin et al., 2020).

DETAILED DESCRIPTION:
Humans are fundamentally social animals. The ability to operate within large social networks requires considerable cognitive capacity, often referred to as social cognition. One social cognitive process thought to involve embodied and nonembodied processes is perspective-taking. Recently, the right temporoparietal junction (rTPJ) has been suggested as a key hub for embodied processing relevant to social cognition. A study of Martin et al. (2020) could further provide causal evidence that the right temporoparietal junction is involved specifically in the embodied component of perspective-taking. Specifically, HD-tDCS (high-definition transcranial direct current stimulation) to the right temporoparietal junction, but not another hub of the social brain (dorsomedial PFC), increased the effect of body position during perspective-taking, but not tracking. As social cognition is affected by the aging process and decline of socio-cognitive abilities is a key feature of neurological diseases such as Alzheimer's or Parkinson's disease, the aim of the present study is to replicate the findings of Martin et al., (2020) in a sample of healthy older adults to better understand the modulation of socio-cognitive processes in older age.

The aim of the study is to explore the effect of transcranial direct current stimulation (tDCS) on either the right tempo-parietal junction (rTPJ) or the dorsomedial prefrontal cortex (dmPFC) in healthy older adults (replication in a different sample of a study by Martin et al., 2020). 60 healthy older adults and 30 younger participants (serving as a control group) will be tested in a Reading the Eyes in the Mind Task (RMET) and a Task of Visual Perspective Taking (VPT) , while stimulation either the rTPJ or the dmPFC with either active or sham tDCS (stimulation only in the group of older participants). In the RMET the expectation is that older participants have higher reaction times after correct answers under rTPJ tDCS. No stimulation effects of the dmPFC are expected. In the VPT older participants are expected to have a selective effect on body position (similar to the results of Martin et al., 2020) under rTPJ stimulation, but not dmPFC stimulation.

A further focus of the study is how functional and structural connectivity of the brain and individual differences measured with an MRI assessment influence with the success of the RMET and VPT paradigms in an explorative research question.

ELIGIBILITY:
Inclusion Criteria:

* healthy older (60 - 80 years) and younger (18 - 30 years) participants
* German as their main language or sufficient german skills to understand the experiment and the task

Exclusion Criteria:

* participants with neuropsychological or psychiatric disease that affect cognition.
* standard MRI exclusion criteria (e.g. pregnancy, metal implants)
* standard tDCS exclusion criteria (e.g. metal implants in the head)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants were asked to name the gender with which they identify.
Enrollment: 90 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Response Time in milliseconds in Visual-Perspective Taking Paradigm (VPT) in the active tDCS. | at Day 1 or 7 (depends on randomization)
  The outcome in the VPT paradigm will be response time in milliseconds (for correct answers only).
Response Time in milliseconds in Visual-Perspective Taking Paradigm (VPT) in the sham tDCS. | at Day 1 or 7 (depends on randomization)
  The outcome in the VPT paradigm will be response time in milliseconds (for correct answers only).
Response Time in milliseconds in the Reading the mind in the eyes test (RMET) in the active tDCS. | at Day 1 or 7 (depends on randomization)
  Outcome in the RMET will be reaction times in milliseconds (of correct answers only) in either rTPJ or dmPFC stimulation in comparison to sham stimulation.
Response Time in milliseconds in the Reading the mind in the eyes test (RMET) in the sham tDCS. | at Day 1 or 7 (depends on randomization)
  Outcome in the RMET will be reaction times in milliseconds (of correct answers only) in either rTPJ or dmPFC stimulation in comparison to sham stimulation.

SECONDARY OUTCOMES:
Functional and structural connectivity (via MRI) | MRI Assessment takes places before participants are stimulated with tDCS at Baseline (Day 1).
  It will be investigated how functional and structural connectivity of the brain and individual differences measured with an MRI assessment influence with the success of the RMET and VPT paradigms in an explorative research question.Structural and functional connectivity will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Meinzer, Dr., Principal Investigator — Universitymedicine Greifswald
Locations (1):
- University Medicine Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin AK, Kessler K, Cooke S, Huang J, Meinzer M. The Right Temporoparietal Junction Is Causally Associated with Embodied Perspective-taking. J Neurosci. 2020 Apr 8;40(15):3089-3095. doi: 10.1523/JNEUROSCI.2637-19.2020. Epub 2020 Mar 4. PMID 32132264
- [Derived] Roheger M, Mader A, Riemann S, Niemann F, Kessler K, Martin AK, Meinzer M. Intact embodiment during perspective-taking in older adults is not affected by focal tDCS. Geroscience. 2025 Dec;47(6):6823-6837. doi: 10.1007/s11357-025-01554-4. Epub 2025 Feb 19. PMID 39966250